CLINICAL TRIAL: NCT02377648
Title: Everolimus-eluting Bioresorbable Vascular Scaffold System in the Treatment of Cardiac Allograft Vasculopathy in Heart Transplant Recipients: A Prospective Multicenter Pilot Study
Brief Title: Safety and Efficacy of Everolimus - Eluting Bioresorbable Vascular Scaffold for Cardiac Allograft Vasculopathy
Acronym: CART
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Flavio Ribichini, Medical Doctor, Universita di Verona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CART
Record Dates: First submitted 2015-02-16; First posted 2015-03-03 (Estimated); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Cardiac Allograft Vasculopathy
Keywords: Cardiac Allograft Vasculopathy; Heart Transplant; Bioresorbable Vascular Scaffold

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABSORB Bioresorbable Vascular Scaffold (Experimental): Everolimus-Eluting Bioresorbable Vascular Scaffold implantation
  Interventions: Device: Everolimus-Eluting Bioresorbable Vascular Scaffold (ABSORB)

INTERVENTIONS:
Device: Everolimus-Eluting Bioresorbable Vascular Scaffold (ABSORB) — Placement of bioresorbable vascular scaffold in presence of at least one critical angiographic de novo lesion (DS ≥70%) or a non-critical angiographic de novo lesion (50% ≤ DS <70%) associated with concomitant signs or symptoms of myocardial ischemia.

SUMMARY:
The CART Pilot study was designed to provide preliminary observations (about performance and safety) and generate hypotheses for future studies . The primary goal of the study is to evaluate the performance at one year of second-generation ABSORB Bioresorbable Vascular Scaffold (BVS)(Abbott Vascular, Santa Clara, CA , USA), the Everolimus Eluting Bioresorbable Vascular Scaffold, in heart transplant recipients affected by cardiac allograft vasculopathy (CAV) and significative coronary stenosis.

The secondary objectives are:

* to collect data about the procedural and clinical outcomes post-procedure , 30 days, 180 days and at 1,2 and 3-year follow-up, of patients who underwent ABSORB BVS implantation in order to investigate the safety of the device in CAV population;
* to evaluate the progression of the disease and the its interactions with the study device by using data derived from multi-imaging invasive techniques.

The vascular reparative therapy and in particular the BVS technology showing important advantages in terms of endothelial preservation, adequate vasomotion, and restoration of the media and adventitia of the vessel wall, could represent a new and more effective therapeutic option, compared to bare-metal and drug-eluting stent technologies, for transplanted patients, since all these mechanisms may, at least in part, counteract the detrimental changes leading to CAV, namely constrictive remodeling and rapid atherosclerosis progression.

Subjects enrolled into the clinical study will be male or female derived from the heart transplant recipients population of every participating center. The clinical study will enroll 30 subjects. Subjects, who underwent the yearly expected coronary angiography follow-up after heart transplant surgery, meeting the general and angiographic inclusion and exclusion criteria (eligibility will be assessed by Heart Team consensus) will be asked to sign an informed consent form. Subjects who do not meet inclusion and exclusion criteria are subject to the standard follow-up of heart transplant (HTx) recipients and will undergo to an invasive evaluation after 365 ± 28 days.

The study comprises two distinct phases:

* the enrollment phase which starts with the recruitment of the first subject and it is planned to last one year;
* the follow-up phase which is planned to last three years from the enrollment of the last patient.

The total duration of the study will be of four years, including both the enrollment and the follow-up phases

ELIGIBILITY:
Inclusion Criteria:

* General Inclusion criteria:

All the enrolled patients must be heart transplanted recipients. The inclusion criteria must follow the most recent instructions for use (IFU) for BVS which may include but are not

Limited to the following:

* Patient must be at least 18 years of age at the time of signing the Informed Consent Form
* Patient must be eligible for percutaneous coronary intervention (PCI)
* Patient is to be treated for de novo lesions located in previously untreated vessels.
* Patient must agree to undergo all required follow-up visits and data collection.

Angiographic inclusion criteria:

• Presence of at least one critical angiographic de novo lesion (DS ≥70%) or a non-critical angiographic de novo lesion (50% ≤ DS <70%) associated with concomitant signs or symptoms of myocardial ischemia. Any intermediate lesion without a clear evidence of ischemia will be interrogated by means of fractional flow reserve assessment with a pressure wire, as recommended by current international guidelines

Exclusion Criteria:

* General Exclusion criteria:

  * Inability to obtain a signed informed consent from potential patient.
  * Contraindications for drug eluting scaffold implantation (known hypersensitivity or contraindication to aspirin, both heparin and bivalirudin, clopidogrel, ticlopidine, prasugrel, and ticagrelor, everolimus, poly (L-lactide), poly (D,L-lactide), or platinum, or with contrast sensitivity, who cannot be adequately premedicated).
  * Female patients with childbearing potential with a positive pregnancy test within 7 days prior to the index procedure.
  * Prior Coronary Artery Bypass Graft (CABG) at any time or planned CABG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Restenosis rate (bioresorbable vascular scaffold), defined as >50% narrowing at the stent site or 5 mm proximal or distal to the stent, as assessed by Quantitative Coronary Analysis. | One Year

SECONDARY OUTCOMES:
Device success (lesion based analysis) | Basal procedure
Procedural success (subject based analysis) | Basal procedure
Death (cardiac, vascular, non-cardiovascular) | 30 days, 180 days, 2 years and 3 years
Myocardial infarction (MI: Q wave Myocardial Infarction (QMI) | 30 days, 180 days, 1 year, 2 years and 3 years
Target lesion revascularization (TLR) | 30 days, 180 days, 1 year, 2 years and 3 years
Target vessel revascularization (TVR) | 30 days, 180 days, 1 year, 2 years and 3 years
Non-target vessel revascularization (NTVR) | 30 days, 180 days, 1 year, 2 years and 3 years
Composite (Death/All MI/ Graft failure) | 30 days, 180 days, 1 year, 2 years and 3 years
Composite (Cardiac death/TV-MI/TLR ) | 30 days, 180 days, 1 year, 2 years and 3 years
Composite (Cardiac death/all MI/TLR ) | 30 days, 180 days, 1 year, 2 years and 3 years
Composite (Cardiac death/all MI/TVR) | 30 days, 180 days, 1 year, 2 years and 3 years
Composite (Death/All MI/all revascularization) | 30 days, 180 days, 1 year, 2 years and 3 years
Scaffold thrombosis | 30 days, 180 days, 1 year, 2 years and 3 years
  Timing (Acute)
Scaffold thrombosis | 30 days, 180 days, 1 year, 2 years and 3 years
  Timing (Subacute)
Scaffold thrombosis | 30 days, 180 days, 1 year, 2 years and 3 years
  Timing (Late)
Scaffold thrombosis | 30 days, 180 days, 1 year, 2 years and 3 years
  Timing (Very late)
Scaffold thrombosis | 30 days, 180 days, 1 year, 2 years and 3 years
  Evidence (Definite)
Scaffold thrombosis | 30 days, 180 days, 1 year, 2 years and 3 years
  Evidence (Probable)
Scaffold thrombosis | 30 days, 180 days, 1 year, 2 years and 3 years
  Evidence (Possible)
Angiographic Endpoints | Basal procedure, 1 year and 3 years
  In-scaffold Reference Vessel Diameter (RVD) (mm)
Angiographic Endpoints | Basal procedure, 1 year and 3 years
  In-scaffold Minimal Lumen Diameter (MLD) (mm)
Angiographic Endpoints | Basal procedure, 1 year and 3 years
  In-scaffold Diameter Stenosis (DS) (%)
Angiographic Endpoints | Basal procedure, 1 year and 3 years
  In-scaffold late loss (mm)
Angiographic Endpoints | Basal procedure, 1 year and 3 years
  Proximal late loss (mm)
Angiographic Endpoints | Basal procedure, 1 year and 3 years
  Distal late loss (mm)
Angiographic Endpoints | Basal procedure, 1 year and 3 years
  In-scaffold absolute minimal luminal area (mm2)
Angiographic Endpoints | Basal procedure, 1 year and 3 years
  In-scaffold minimal luminal cross sectional area (mm2)
Angiographic Endpoints | Basal procedure, 1 year and 3 years
  In-segment late loss (mm) In-stent binary restenosis (%)
Angiographic Endpoints | Basal procedure, 1 year and 3 years
  In-segment binary restenosis
Intravascular Ultrasound/Intravascular Ultrasound-Virtual Histology Endpoints | Basal procedure and 3 years
  Vessel (EEM) area (mm2)
Intravascular Ultrasound/Intravascular Ultrasound-Virtual Histology Endpoints | Basal procedure and 3 years
  Vessel volume (mm3)
Intravascular Ultrasound/Intravascular Ultrasound-Virtual Histology Endpoints | Basal procedure and 3 years
  Average lumen area (mm2)
Intravascular Ultrasound/Intravascular Ultrasound-Virtual Histology Endpoints | Basal procedure and 3 years
  Lumen volume (mm3)
Intravascular Ultrasound/Intravascular Ultrasound-Virtual Histology Endpoints | Basal procedure and 3 years
  Plaque area (mm2)
Intravascular Ultrasound/Intravascular Ultrasound-Virtual Histology Endpoints | Basal procedure and 3 years
  Plaque volume (mm3)
Intravascular Ultrasound/Intravascular Ultrasound-Virtual Histology Endpoints | Basal procedure and 3 years
  Minimal lumen area (mm2)
Intravascular Ultrasound/Intravascular Ultrasound-Virtual Histology Endpoints | Basal procedure and 3 years
  Lumen area stenosis (%)
Intravascular Ultrasound/Intravascular Ultrasound-Virtual Histology Endpoints | Basal procedure and 3 years
  Vessel volume index (mm3/mm)
Intravascular Ultrasound/Intravascular Ultrasound-Virtual Histology Endpoints | Basal procedure and 3 years
  Lumen volume index (mm3/mm)
Intravascular Ultrasound/Intravascular Ultrasound-Virtual Histology Endpoints | Basal procedure and 3 years
  Plaque volume index (mm3/mm)
Intravascular Ultrasound/Intravascular Ultrasound-Virtual Histology Endpoints | Basal procedure and 3 years
  Plaque burden, %
Intravascular Ultrasound/Intravascular Ultrasound-Virtual Histology Endpoints | Basal procedure and 3 years
  Projected MLD (mm)
Intravascular Ultrasound/Intravascular Ultrasound-Virtual Histology Endpoints | Basal procedure and 3 years
  Dense calcium volume, area, percentage
Intravascular Ultrasound/Intravascular Ultrasound-Virtual Histology Endpoints | Basal procedure and 3 years
  Necrotic core volume, area, percentage
Intravascular Ultrasound/Intravascular Ultrasound-Virtual Histology Endpoints | Basal procedure and 3 years
  Fibrofatty volume, area, percentage
Intravascular Ultrasound/Intravascular Ultrasound-Virtual Histology Endpoints | Basal procedure and 3 years
  Fibrous volume, area, percentage
Optical Coherence Tomography Endpoints | Basal procedure and 3 years
  Maximal intimal thickness (MIT) (mm)
Optical Coherence Tomography Endpoints | Basal procedure and 3 years
  Media thickness at MIT (mm)
Optical Coherence Tomography Endpoints | Basal procedure and 3 years
  Mean lumen area (mm2)
Optical Coherence Tomography Endpoints | Basal procedure and 3 years
  Intimal area (mm2)
Optical Coherence Tomography Endpoints | Basal procedure and 3 years
  Maximal, minimal and mean lumen diameter (mm)
Optical Coherence Tomography Endpoints | Basal procedure and 3 years
  Discernible struts
Optical Coherence Tomography Endpoints | Basal procedure and 3 years
  Atherosclerosis assessment (Eccentric plaque)
Optical Coherence Tomography Endpoints | Basal procedure and 3 years
  Atherosclerosis assessment (Calcification)
Optical Coherence Tomography Endpoints | Basal procedure and 3 years
  Atherosclerosis assessment (Lipid)
Optical Coherence Tomography Endpoints | Basal procedure and 3 years
  Vulnerable plaque assessment (thin-cap fibroatheroma)
Optical Coherence Tomography Endpoints | Basal procedure and 3 years
  Vulnerable plaque assessment (macrophages)
Optical Coherence Tomography Endpoints | Basal procedure and 3 years
  Vulnerable plaque assessment (microchannels)
Optical Coherence Tomography Endpoints | Basal procedure and 3 years
  Vulnerable plaque assessment (calcific nod)
Optical Coherence Tomography Endpoints | Basal procedure and 3 years
  Lesions assessment (Intimal laceration)
Optical Coherence Tomography Endpoints | Basal procedure and 3 years
  Lesions assessment (plaque rupture)
Optical Coherence Tomography Endpoints | Basal procedure and 3 years
  Lesions assessment (intraluminal thrombus)
Optical Coherence Tomography Endpoints | Basal procedure and 3 years
  Lesions assessment (layered complex plaque)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio L Ribichini, MD, Principal Investigator — Universita di Verona; Michele Pighi, MD, Principal Investigator — Universita di Verona
Locations (10):
- Italy (8):
  - Azienda Ospedaliera Brotzu, Cagliari
  - Azienda Ospedaliera Specialistica Dei Colli, Naples
  - Azienda Ospedaliera Di Padova, Padua
  - Fondazione Irccs Policlinico San Matteo, Pavia
  - Azienda Ospedaliera San Camillo Forlanini, Rome
  - European Hospital, Rome
  - Azienda Sanitaria Universitaria Integrata Di Udine (Asuiud), Udine
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Netherlands (2):
  - Cardialysis Core Laboratory For Imaging, Rotterdam
  - Thoraxcenter, Universtity of Rotterdam, Rotterdam

REFERENCES:
- [Background] Ribichini F, Pighi M, Faggian G, Vassanelli C. Bioresorbable vascular scaffolds in cardiac allograft vasculopathy: a new therapeutic option. Am J Med. 2013 Nov;126(11):e11-4. doi: 10.1016/j.amjmed.2013.05.025. No abstract available. PMID 24157291
- [Background] Authors/Task Force members; Windecker S, Kolh P, Alfonso F, Collet JP, Cremer J, Falk V, Filippatos G, Hamm C, Head SJ, Juni P, Kappetein AP, Kastrati A, Knuuti J, Landmesser U, Laufer G, Neumann FJ, Richter DJ, Schauerte P, Sousa Uva M, Stefanini GG, Taggart DP, Torracca L, Valgimigli M, Wijns W, Witkowski A. 2014 ESC/EACTS Guidelines on myocardial revascularization: The Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS)Developed with the special contribution of the European Association of Percutaneous Cardiovascular Interventions (EAPCI). Eur Heart J. 2014 Oct 1;35(37):2541-619. doi: 10.1093/eurheartj/ehu278. Epub 2014 Aug 29. No abstract available. PMID 25173339
- [Background] Taylor DO, Edwards LB, Aurora P, Christie JD, Dobbels F, Kirk R, Rahmel AO, Kucheryavaya AY, Hertz MI. Registry of the International Society for Heart and Lung Transplantation: twenty-fifth official adult heart transplant report--2008. J Heart Lung Transplant. 2008 Sep;27(9):943-56. doi: 10.1016/j.healun.2008.06.017. No abstract available. PMID 18765186
- [Background] Tomai F, Adorisio R, De Luca L, Pilati M, Petrolini A, Ghini AS, Parisi F, Pongiglione G, Gagliardi MG. Coronary plaque composition assessed by intravascular ultrasound virtual histology: association with long-term clinical outcomes after heart transplantation in young adult recipients. Catheter Cardiovasc Interv. 2014 Jan 1;83(1):70-7. doi: 10.1002/ccd.25054. Epub 2013 Jul 16. PMID 23765788
- [Background] Serruys PW, Ormiston JA, Onuma Y, Regar E, Gonzalo N, Garcia-Garcia HM, Nieman K, Bruining N, Dorange C, Miquel-Hebert K, Veldhof S, Webster M, Thuesen L, Dudek D. A bioabsorbable everolimus-eluting coronary stent system (ABSORB): 2-year outcomes and results from multiple imaging methods. Lancet. 2009 Mar 14;373(9667):897-910. doi: 10.1016/S0140-6736(09)60325-1. PMID 19286089
- [Derived] Pighi M, Tomai F, Petrolini A, de Luca L, Tarantini G, Barioli A, Colombo P, Klugmann S, Ferlini M, Ormezzano MF, Loi B, Calabro P, Bianchi RM, Faggian G, Forni A, Vassanelli C, Valgimigli M, Ribichini F. Everolimus-Eluting Bioresorbable Vascular Scaffold System in the Treatment of Cardiac Allograft Vasculopathy: the CART (Cardiac Allograft Reparative Therapy) Prospective Multicenter Pilot Study. J Cardiovasc Transl Res. 2016 Feb;9(1):40-8. doi: 10.1007/s12265-015-9665-x. Epub 2015 Dec 18. PMID 26684009